CLINICAL TRIAL: NCT00266006
Title: Safety of Eptacog Alfa (Activated) (Genetical Recombination) on Adverse Events and Serious Adverse Events in Patients With Acute Intracerebral Haemorrhage.
Brief Title: Factor VIIa in Acute Intracerebral Haemorrhage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: F7ICH-1602; JapicCTI-050194 (Registry Identifier: japic)
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Acquired Bleeding Disorder; Intracerebral Haemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Factor VII

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: eptacog alfa (activated)
  Other Names: activated recombinant human factor VII

SUMMARY:
This trial is conducted in Japan. The purpose of this trial is to evaluate the safety and preliminary efficacy of Activated Recombinant Factor VII (NN-007) in patients with acute intracerebral haemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous ICH

Exclusion Criteria:

* Time of ICH onset > 3 hours
* Patients with secondary ICH
* Pre-existing disability
* Hemophilia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The Occurrence of thromboembolic serious adverse event | Until 90 days

SECONDARY OUTCOMES:
Reducing disability and improving clinical outcome
Reducing haematoma growth

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com